CLINICAL TRIAL: NCT06316141
Title: Effects of Aquatic vs Land Based Jogging on BMI, Cardiorespiratory Endurance and QoL in Overweight Adults
Brief Title: Effects of Aquatic vs Land Based Jogging in Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0352
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Overweight
Keywords: Aqua jogging; Endurance; Hydrotherapy; Land jogging; Overweight; Quality of Life
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (Experimental): Aqua Jogging Group
  Interventions: Other: Aqua Jogging
- Experimental Group B (Experimental): Land based Jogging Group
  Interventions: Other: Land based Jogging

INTERVENTIONS:
Other: Aqua Jogging — This group performed aqua jogging for 60 minutes consisting of 10 minutes warming up, 40 minutes aqua jogging or land jogging and 10 minutes cooling down.
  Arms: Experimental Group A
Other: Land based Jogging — This group performs land jogging for 60 minutes consisting of 10 minutes warming up, 40 minutes aqua jogging or land jogging and 10 minutes cooling down.
  Arms: Experimental Group B

SUMMARY:
Obesity raises the risk of chronic illnesses in adults, especially heart disease, type II diabetes, and osteoarthritis. One way to combat obesity is by physical activity, and water-based exercise (hydrotherapy) is recognized as an enhancement of the more common on land physical activity. Obesity is associated with several negative health outcomes, including cardiovascular disease (CVD), cardiac enlargement, gallbladder disease, diabetes, several cancers, osteoarthritis, and sleeping disorders .In addition to being a significant predictor of coronary heart disease and heart failure. obesity is indirectly related to cardiovascular health through its association with several other CVD risk factors, including hypertension, high cholesterol, low high-density lipoprotein (HDL) cholesterol, high triglycerides, and diabetes Therefore, obesity is a primary target for interventions to decrease overall cardiovascular risk. It is a randomized clinical trial conducted at the University OF Central Punjab Lahore. Convenience sampling technique will be used .Participants will be recruited through simple random sampling by sealed opaque envelope method into two Groups .Group A and Group B. Group A:Aqua jogging group: This group will perform aqua jogging for 60 minutes consisting of 10 minutes warming up, 40 minutes aqua jogging or land jogging and 10 minutes cooling down. Group B: Land based jogging group: This group will perform land jogging for 60 minutes consisting of 10 minutes warming up, 40 minutes aqua jogging or land jogging and 10 minutes cooling down. Assessment tools for this study will be cooper's 1.5 miles run test for cardiorespiratory endurance and health related quality of life questionnaire for Quality of life. The study will be completed within 10 months after synopsis approval from ethical Committee of RCRS & AHS .Data will be entered and analysed by SPSS version 25. After assessing the normality of data, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Exclusion Criteria:

* Individuals having exercise induced asthma
* Any skin disease- open wound infection
* Participants having hydrophobia
* Individuals with chronic issues & physical defects
* Participants with cognitive impairments
* Ongoing medications that would be of lipid metabolism, menstruation, history of gastrointestinal infection

Inclusion Criteria:

* BMI: 25 - 30 kg/m2
* Gender: both
* Age: 20-59 years

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Endurance(cooper; s1.5 miles run) | 12 weeks
  Cardiorespiratory endurance measured by Cooper tests an easy running test of .cardiorespiratory endurance is the 2.4 km (1.5 mile) run test, which simply needs a timer and a running track. The test's objective is to cover the 2.4 km course in the quickest amount of time feasible. All competitors are positioned in a starting line formation. The clock starts when they are told to "go," and they then start running at their own pace. It determines the amount of cardiovascular fitness by estimating the body's capacity to transport oxygen. Pre-Post Readings will be taken
Quality of life (health related QOL SF 36 Questionnaire) | 12 weeks
  The Short Form Survey (SF-36) is a tool used to measure various aspects of quality of life, such as body pain, physical well-being or functionality. Restrictions on role performance brought on by issues with one's physical, mental, or social well-being as well as one's general sense of health. Pre-post readings will be taken
BMI | 12 weeks
  Measurement for BMI will perform by dividing a person's weight in kilograms by the square of height in meters .in which Height will be measured using an inches tape with participants on bare feet. Weight measurement will be taken by weighing machine. A high BMI can indicate high body fatness. Pre-post Readings will be taken12

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Muriam Ghani, MSCPPT, Principal Investigator — Ripha International University-LHR
Locations (1):
- University of Central Punjab (sports complex) Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sturm R, Hattori A. Morbid obesity rates continue to rise rapidly in the United States. Int J Obes (Lond). 2013 Jun;37(6):889-91. doi: 10.1038/ijo.2012.159. PMID 22986681
- [Background] Lee BA, Oh DJ. The effects of aquatic exercise on body composition, physical fitness, and vascular compliance of obese elementary students. J Exerc Rehabil. 2014 Jun 30;10(3):184-90. doi: 10.12965/jer.140115. eCollection 2014 Jun. PMID 25061599
- [Background] Czernichow S, Kengne AP, Stamatakis E, Hamer M, Batty GD. Body mass index, waist circumference and waist-hip ratio: which is the better discriminator of cardiovascular disease mortality risk?: evidence from an individual-participant meta-analysis of 82 864 participants from nine cohort studies. Obes Rev. 2011 Sep;12(9):680-7. doi: 10.1111/j.1467-789X.2011.00879.x. Epub 2011 Apr 27. PMID 21521449
- [Background] Lehnert T, Sonntag D, Konnopka A, Riedel-Heller S, Konig HH. Economic costs of overweight and obesity. Best Pract Res Clin Endocrinol Metab. 2013 Apr;27(2):105-15. doi: 10.1016/j.beem.2013.01.002. Epub 2013 Feb 28. PMID 23731873
- [Background] Savoye M, Shaw M, Dziura J, Tamborlane WV, Rose P, Guandalini C, Goldberg-Gell R, Burgert TS, Cali AM, Weiss R, Caprio S. Effects of a weight management program on body composition and metabolic parameters in overweight children: a randomized controlled trial. JAMA. 2007 Jun 27;297(24):2697-704. doi: 10.1001/jama.297.24.2697. PMID 17595270
- [Background] Volaco A, Cavalcanti AM, Filho RP, Precoma DB. Socioeconomic Status: The Missing Link Between Obesity and Diabetes Mellitus? Curr Diabetes Rev. 2018;14(4):321-326. doi: 10.2174/1573399813666170621123227. PMID 28637406
- [Background] Aballay LR, Eynard AR, Diaz Mdel P, Navarro A, Munoz SE. Overweight and obesity: a review of their relationship to metabolic syndrome, cardiovascular disease, and cancer in South America. Nutr Rev. 2013 Mar;71(3):168-79. doi: 10.1111/j.1753-4887.2012.00533.x. Epub 2013 Jan 7. PMID 23452284